CLINICAL TRIAL: NCT06551649
Title: Contrasting Chronic Inflammation and Neurodegeneration Using the Human Amniotic Mesenchymal Cell Secretome as an Innovative Therapeutic Strategy
Brief Title: Human Amniotic Mesenchymal Cell Secretome for Neurodegeneration and Neuroinflammation
Acronym: CONTRASTOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6823
Record Dates: First submitted 2024-07-16; First posted 2024-08-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients diagnosed with amyotrophic lateral sclerosis (Experimental): Amyotrophic lateral sclerosis patients will be recruited to obtain venous blood draw and skin biopsy, to optimize a three-dimensional cellular model of multiple sclerosis in which determine the neuroprotective and anti-inflammatory/immunomodulatory effects of the human amniotic mesenchymal stromal cell secretome.
  Interventions: Other: Venous blood draw and skin biopsy
- Patients diagnosed with multiple sclerosis (Experimental): Multiple sclerosis patients will be recruited to obtain venous blood draw and skin biopsy, to optimize a three-dimensional cellular model of multiple sclerosis in which determine the neuroprotective and anti-inflammatory/immunomodulatory effects of the human amniotic mesenchymal stromal cell secretome.
  Interventions: Other: Venous blood draw and skin biopsy
- Healthy volunteers, patients' unaffected spouses (Active Comparator): Spouses of patients will be enrolled as healthy controls, matching their age and male-to-female ratio for both conditions, to obtain venous blood draw and skin biopsy, in order to develop a control model against which to evaluate the preclinical efficacy of the human amniotic mesenchymal stromal cell secretome.
  Interventions: Other: Venous blood draw and skin biopsy

INTERVENTIONS:
Other: Venous blood draw and skin biopsy — The skin tissue will be used to isolate fibroblasts, which will then be reprogrammed into induced pluripotent stem cells (iPSCs). These iPSCs will be differentiated to develop patient-specific and control organoids. The blood samples will be used to isolate peripheral blood mononuclear cells (PBMC) to study the contribution of inflammation in the in vitro models developed.

SUMMARY:
Neurodegenerative diseases are debilitating conditions characterized by chronic inflammation, leading to dysfunction of both the non-neuronal cellular components of the central nervous system and peripheral blood immune cells. Thus, it is crucial to develop an innovative therapeutic strategy that not only effectively contrast neurodegeneration but also aims to reduce inflammation.

The overall aim of the study is to provide a preclinical in vitro demonstration of the immunomodulatory and pro-regenerative potential of the human amniotic mesenchymal stromal cell (hAMSC) secretome in counteracting neurodegeneration.

This potential will be evaluated in three-dimensional in vitro models of neurodegenerative diseases, such as amyotrophic lateral sclerosis (ALS) and chronic demyelinating disease (multiple sclerosis - MS). To this end, the study includes sample collection from patients without pharmacological treatment and without medical devices. Patients diagnosed with ALS, patients diagnosed with MS, and healthy volunteers will be recruited to collect blood samples and skin biopsies. Patient-specific and control organoid platforms, mimicking cellular heterogeneity and tridimensional interactions within the central nervous system including the inflammatory compartment, will be developed to be used as a valuable tool to investigate the in vitro efficacy of the hAMSC secretome.

ELIGIBILITY:
Inclusion Criteria:

* For patients with amyotrophic lateral sclerosis (ALS): aged between 50 and 60 years and similar age of onset and duration of the disease.
* For patients with multiple sclerosis (MS): with recently confirmed diagnosis of MS, aged between 20 and 50 years and considering the male-to-female ratio in MS of approximately 2:1.
* For healthy volunteers: spouses of patients unaffected by any neurological disease and matching their age and gender ratio for both conditions.

Exclusion Criteria:

* Patients who do not consent to participate in the study.
* MS patients who have received treatment with immunomodulators or corticosteroids and are in an acute phase of the disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Neurite length measurement in a three-dimensional cellular model of amyotrophic lateral sclerosis. | 18 months
  Organoids from induced pluripotent stem cells (iPSCs) isolated from skin biopsies of 6 amyotrophic lateral sclerosis (ALS) patients and 6 healthy controls will be generated. Neurite degeneration will be measured in fluorescence microscopy as total βIII-TUBULIN-positive fiber length divided by the number of βIII-TUBULIN-positive cells in micrometers. Measurements will be taken from at least 5 ALS and 5 control organoids to analyze correlations and differences between groups. The significance level for statistical tests and models is set at 0.05.
Percentage of apoptotic cells in a three-dimensional cellular model of amyotrophic lateral sclerosis. | 18 months
  Organoids from induced pluripotent stem cells (iPSCs) isolated from skin biopsies of 6 amyotrophic lateral sclerosis (ALS) patients and 6 healthy controls will be generated. Apoptosis will be assessed by the percentage of propidium iodide-positive cells, representing the proportion of dead cells relative to the total number of cells. Measurements will be taken from at least 5 ALS and 5 control organoids to analyze correlations and differences between groups. The significance level for statistical tests and models is set at 0.05.
Area measurement of damaged myelin in a three-dimensional cellular model of multiple sclerosis. | 18 months
  Organoids from induced pluripotent stem cells (iPSCs) isolated from skin biopsies of 6 multiple sclerosis (MS) patients and 6 healthy controls will be generated. Myelin sheath damage will be assessed via immunofluorescence as the reduction in myelin marker-stained area versus total section area. Measurements will be taken from at least 5 MS and 5 control organoids to analyze correlations and differences between groups. The significance level for statistical tests and models is set at 0.05.
Number of inflamed microglial cells in a three-dimensional cellular model of multiple sclerosis. | 18 months
  Organoids from induced pluripotent stem cells (iPSCs) isolated from skin biopsies of 6 multiple sclerosis (MS) patients and 6 healthy controls will be generated. Microglial activation will be assessed by morphological variations, classifying cells as homeostatic, ramified, hyper-ramified, or amoeboid. Inflammatory microglia increase will be defined as the proportion of activated morphology cells relative to total cell count. Inflammatory markers HLA-DR and iNOS will be evaluated in terms of CD68 and IBA1 positive cells and fluorescence intensity. Measurements will be taken from at least 5 MS and 5 control organoids to analyze correlations and differences between groups. The significance level for statistical tests and models is set at 0.05.
Neurite length measurement in amyotrophic lateral sclerosis organoids after treatment with human amniotic mesenchymal stromal cell secretome. | 24 months
  Neurite length in amyotrophic lateral sclerosis (ALS)-derived organoids treated with human amniotic mesenchymal stromal cell (hAMSC) secretome will be quantified using fluorescence microscopy as the total βIII-TUBULIN-positive fiber length divided by the number of βIII-TUBULIN-positive cells. The ability of the hAMSC secretome to restore ALS organoids (at least 5) to values close to healthy-donors organoids (at least 5) will be evaluated. The significance level is set at 0.05.
Percentage of apoptotic cells in amyotrophic lateral sclerosis organoids after treatment with human amniotic mesenchymal stromal cell secretome. | 24 months
  Apoptosis will be measured by the reduction in propidium iodide-positive cells, expressed as a percentage of the total cells, in amyotrophic lateral sclerosis (ALS)-derived organoids treated with human amniotic mesenchymal stromal cell (hAMSC) secretome. The ability of the hAMSC secretome to restore ALS organoids (at least 5) to values close to healthy-donors organoids (at least 5) will be evaluated. The significance level is set at 0.05.
Area measurement of damaged myelin in multiple sclerosis organoids after treatment with human amniotic mesenchymal stromal cell secretome. | 24 months
  Reduction of demyelinated areas in multiple sclerosis (MS)-derived organoids treated with human amniotic mesenchymal stromal cell (hAMSC) secretome will be measured by the increase in mature oligodendrocyte markers relative to total section area. The ability of the hAMSC secretome to restore MS organoids (at least 5) to values close to healthy-donors organoids (at least 5) will be evaluated. The significance level is set at 0.05.
Number of immunoregulatory microglial cells in multiple sclerosis organoids after treatment with human amniotic mesenchymal stromal cell secretome. | 24 months
  The acquisition of an immunoregulatory phenotype will be determined in multiple sclerosis (MS)-derived organoids after treatment with human amniotic mesenchymal stromal cell (hAMSC) secretome by analyzing cells that are iNOS-negative, Arginase-positive, and HLA-DR low. Immunofluorescence analysis will count the number of cells positive for inflammatory/immunoregulatory markers out of total microglial IBA1+ cells. Fluorescence intensity changes will also be evaluated. The ability of the hAMSC secretome to restore MS organoids (at least 5) to values close to healthy-donors organoids (at least 5) will be evaluated. The significance level is set at 0.05.

SECONDARY OUTCOMES:
Percentage of altered immune phenotypic markers in amyotrophic lateral sclerosis and multiple sclerosis patients | 18 months
  The altered immune phenotype of peripheral blood mononuclear cells (PBMC) from patients with amyotrophic lateral sclerosis (ALS, n=15) and multiple sclerosis (MS, n=15) will be compared to age- and gender-matched healthy controls PBMC (n=30). Flow cytometry will be used to identify alteration in T and B lymphocytes, and monocytes and their subsets, including naïve and memory subsets, senescence status, expression of activation markers, and costimulatory molecules. The percentage of more than 40 markers will be considered and positive expression for each marker will be recorded. Immunophenotypic variation between patient PBMC and healthy control PBMC will be considered statistically significant with a p value < 0,05.

CONTACTS AND LOCATIONS:
Overall Officials: Ornella Parolini, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome